CLINICAL TRIAL: NCT00002023
Title: An Oral Dose-Ranging Finding Study in Patients With HIV Disease, CDC Classification Groups IIB, III, and IV-C2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glaxo Wellcome (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 014C; 013
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1995-02

CONDITIONS: HIV Infections
Keywords: Dose-Response Relationship, Drug; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Zidovudine
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Zidovudine

INTERVENTIONS:
Drug: Zidovudine

SUMMARY:
To establish the relationship between the oral dose of zidovudine (AZT) and its hematologic toxicity. AZT has preliminarily been shown to decrease significant events and death in a group of AIDS / Pneumocystis carinii pneumonia (PCP) and AIDS related complex (ARC) patients followed at this time for a limited period. If these data withstand further follow-up, it appears that AZT is a potential antiretroviral agent that may have application in the use of all stages of HIV disease. At this time the optimal dose that will not cause significant toxicity is not known. If this drug has widespread application, it becomes imperative to further study both the dose and the toxicity. Patients with documented HIV viremia and who are well will be evaluated in a dose-escalating protocol for toxicity, persistent viremia, evidence of improvement of immune dysfunction, and the development of further manifestation of HIV disease. Drug levels will be monitored and correlated with the toxicity and viremia.

ELIGIBILITY:
Inclusion Criteria

Patients must have HIV reactivity.

* Patients must belong to one of the following three groups according to the CDC classification:
* IIB - including only those patients with autoimmune thrombocytopenia (platelet count = or < 100000 platelets/mm3).
* OR Lymphopenia (lymphocyte count = or < 1000 cells/mm3).
* OR Helper cell lymphopenia (helper cells < the mean of normals).
* OR CDC classification III or IV-C2.
* Patients with = or < involuntary 10 percent weight loss in the last 6 months.
* ECOG performance status 0 or 1.
* Weigh 70 kg + or - 15 kg in order to standardize the g/kg dosing.
* Positive antibody for HIV by an ELISA test kit. If the ELISA is negative, then eligibility will be confirmed by second confirmatory test, i.e., immunoblot.

Exclusion Criteria

Co-existing Condition:

Patients with the following are excluded:

* AIDS or the CDC classification stage IV except stage IV-C2.
* HIV antibody negative by immunoblot.
* Persistent fevers of > 38.5 degrees C.
* Persistent diarrhea undiagnosed > 1 month.
* Involuntary weight loss of > 10 percent in the 6 months prior to study entry.
* ECOG performance status of 2, 3, or 4.
* Class IV-C2 with prior history of:
* Multidermal herpes zoster.
* Oral candidiasis on more than one occasion.
* Tuberculosis.

Concurrent Medication:

Excluded:

* Other antiretroviral agents.
* Active immunomodulating agents.
* Any other experimental therapy.
* Drugs which cause anemia or neutropenia.
* Drugs which are glucuronidated and may interfere with the metabolism of AZT, i.e., acetaminophen > 5 days.
* Acyclovir systemically administered > 5 days.
* Any other experimental agents.

Patients with the following are excluded:

* AIDS or the CDC classification stage IV except stage IV-C2.
* HIV antibody negative by immunoblot.
* Persistent fevers of > 38.5 degrees C.
* Persistent diarrhea undiagnosed > 1 month.
* Involuntary weight loss of > 10 percent in the 6 months prior to study entry.
* ECOG performance status of 2, 3, or 4.
* Class IV-C2 with prior history of:
* Multidermal herpes zoster.
* Oral candidiasis on more than one occasion.
* Tuberculosis.

Prior Medication:

Excluded within 3 months of study entry:

* Other antiretroviral agents. Active immunomodulating agents.
* Excluded within 2 weeks of study entry:
* Drugs which cause anemia or neutropenia.
* Drugs which are glucuronidated and may interfere with the metabolism of zidovudine (AZT), i.e., acetaminophen > 5 days.
* Acyclovir systemically administered > 5 days.
* Any other experimental agents.

Known active drug abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Glaxo Wellcome Inc, Research Triangle Park, North Carolina, United States